CLINICAL TRIAL: NCT00658736
Title: A Randomized, Triple-Blinded Study of Endoscopic Ultrasound Guided Celiac Plexus Blockade (EUS-CPB) With Bupivicaine and Triamcinolone vs. Bupivicaine Alone for the Treatment of Pain in Chronic Pancreatitis
Brief Title: Efficacy of EUS-guided Celiac Plexus Blockade in Chronic Pancreatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Principal Investigator, Tyler Stevens, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCF IRB 07-729
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): EUS guided celiac block with bupivicaine and triamcinolone. Patient will undergo endoscopic ultrasound and celiac plexus blockade using an EUS needle inserted into the celiac plexus. 20 cc of injectate will be administered.
  Interventions: Drug: Triamcinolone
- 2 (Placebo Comparator): EUS guided celiac block with bupivicaine only. Patient will undergo endoscopic ultrasound and celiac plexus blockade using an EUS needle inserted into the celiac plexus. 20 cc of injectate will be administered.
  Interventions: Drug: Bupivicaine alone

INTERVENTIONS:
Drug: Triamcinolone — Injection of bupivacaine and triamcinolone
  Arms: 1
Drug: Bupivicaine alone — Injection of bupivacaine
  Arms: 2

SUMMARY:
This is a triple-blind, parallel group, randomized controlled trial to assess the benefit of triamcinolone injection as a therapeutic measure for control of chronic pancreatitis pain. The treatment group will undergo EUS-CPB with bupivicaine plus triamcinolone ("therapeutic block"). There control group will undergo EUS-CPB with bupivicaine alone ("diagnostic block").

DETAILED DESCRIPTION:
There are few effective options for the treatment of abdominal pain in chronic pancreatitis. For the past 20 years, percutaneous injection of anesthetic agents into the celiac plexus (celiac plexus blockade or CPB) has been performed by pain anesthesiologists to diagnose the origin of pancreatic pain (visceral vs. non-visceral). Anesthetic blocks provide very short-term and variable pain relief. More recently, endoscopic ultrasound has been used to provide a transgastric approach to the celiac plexus (EUS-CPB).

Corticosteroids may lengthen the effect of CPB to provide longer-lasting pain relief ("therapeutic block"). Case-series report that about 50% of patients experience partial or complete relief lasting an average of 1-2 months. Combined corticosteroid (triamcinolone) and anesthetic (bupivicaine) has now become standard practice for EUS-CPB. However, there have been no randomized controlled trials to prove that corticosteroid blocks are truly therapeutic (i.e. that they lengthen the effect of the typical "diagnostic" CPB with anesthetics). Randomized controlled trials are needed to demonstrate the therapeutic efficacy of CPB with corticosteroids.

This is a triple-blind, parallel group, randomized controlled trial to assess the benefit of triamcinolone injection as a therapeutic measure for control of chronic pancreatitis pain. The treatment group will undergo EUS-CPB with bupivicaine plus triamcinolone ("therapeutic block"). There control group will undergo EUS-CPB with bupivicaine alone ("diagnostic block").

Eligible patients with abdominal pain undergoing EUS for the diagnosis of chronic pancreatitis or EUS-CPB for pancreatic pain will be recruited. Patients will complete a 2-week run-in period to establish baseline pain scores and opioid consumption. Following the run-in, EUS will be performed. If EUS reveals CP (>4 criteria), patients will be randomized to one of the two treatment groups. 74 patients will be randomized and followed for 2 months after the EUS-CPB. The primary endpoint is an improvement in the pain disability index (PDI) of greater than 10 points at 1 month. Secondary endpoints include opioid consumption, duration of pain relief, and quality of life (SF-12).

If this trial shows that the addition of triamcinolone produces a long-lasting (1-month) benefit, then EUS-CPB can be more strongly advocated as a therapeutic option to patients with chronic pancreatitis. If triamcinolone does not produce a benefit over a diagnostic block, then EUS-CPB should be considered a primarily diagnostic measure for differentiation of visceral from non-visceral pain.

ELIGIBILITY:
Inclusion criteria include:

* Age >18 yrs
* Ability for informed consent
* Chronic pancreatic-type abdominal pain (type B) (11).

Exclusion criteria include:

* Pregnancy
* Malignancy
* Recent acute pancreatitis (within 2 months)
* Elevated INR (>1.5) or low platelet count (<75 cells/mm3)
* Allergy to eggs or "caine" anesthetics or corticosteroids; AND
* Becks depression score>20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivicaine Alone: EUS-guided celiac plexus block administered with 20cc Bupivicaine 0.25% solution.
- Bupivicaine Plus Triamcinolone: EUS-guided celiac plexus block administered with 20cc Bupivicaine 0.25% solution mixed with 80 mg Triamcinolone.
Period: Overall Study
Arm/Group | Bupivicaine Alone | Bupivicaine Plus Triamcinolone
Started | 19 | 21
Completed | 13 | 19
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Bupivicaine and Triamcinolone: EUS guided celiac block with bupivicaine and triamcinolone
  Triamcinolone
- Bupivicaine Alone: EUS guided celiac block with bupivicaine only
  Bupivicaine alone
- Total: Total of all reporting groups
Arm/Group | Bupivicaine and Triamcinolone | Bupivicaine Alone | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.9) | 44.1 (12.5) | 41.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 12 | 10 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Disability Index
Description: The Pain Disability Index (PDI) measures patients' responses of the extent to which pain limits their abilities to carry out everyday tasks. The index is scored from 0 (no limitation) to 70 (severe limitation). A decrease in score of 10 points or more is regarded as indicating significant improvement in the ability to carry out daily activities.
Time Frame: 1 month after block
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivicaine and Triamcinolone | Bupivicaine Alone
Number analyzed (Participants) | 21 | 19
Participants | 3 | 3

2. Secondary Outcome: Change From Baseline in Quality of Life Score at 1 Month - SF12 Physical Component
Description: The SF12 survey measures patients' impressions of their level of health and well-being. The results are reported as two scores: A physical component and a mental component, each of which is reported on a scale of 0 (lowest level of health) to 100 (excellent health). Scores that increase from baseline indicate an improvement in patients' feelings of well-being.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivicaine and Triamcinolone | Bupivicaine Alone
Number analyzed (Participants) | 21 | 19
units on a scale | -0.2 (7.5) | 1.7 (8.8)

ADVERSE EVENTS:
Arm/Group | Bupivicaine and Triamcinolone | Bupivicaine Alone
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 4/21 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivicaine and Triamcinolone (N=21) | Bupivicaine Alone (N=19)
Hypertension urgency (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastric hematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes